CLINICAL TRIAL: NCT02614625
Title: A Prospective, Comparative, Observational Study on Spectral-domain Optical Coherence Tomography of the Eye
Brief Title: Spectral-domain Optical Coherence Tomography of the Eye
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Sponsor
Other Study IDs: OCTComparisonstudy1.1
Record Dates: First submitted 2015-10-12; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Cornea; Retina; Refractive Surgery; Macular Edema; Diabetes; Diabetic Macular Edema
MeSH Terms: conditions — Corneal Diseases; Macular Edema; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Normal subjects: Patient with healthy, normal eyes
- Eyes with corneal disease: Subjects that have any of the following conditions
  * Corneal dystrophy or degeneration
  * Corneal scarring
  * Corneal ulcer
  * Corneal injury
  * Keratoconus
  * Patients who had undergone corneal surgery
  * Patients with other corneal disease
- Eyes with retinal disease: Subjects that have any of the following conditions:
  * Diabetic macular edema
  * Cystoid macular edema
  * Age related macular degeneration
  * Retinal vascular disorders (e.g. retinal artery occlusion)
  * Epiretinal membrane
  * Choroidal nevus
  * Macular hole
  * Patients who had undergone retinal surgery
  * Patients with other retinal disease
- Eyes with glaucoma: Eyes diagnosed with glaucoma of any type and any stage

SUMMARY:
An increasing number of clinical studies on SD-OCT of ocular pathologies and potential new clinical applications has recently been published in the peer-reviewed literature. However, the successful use of SD-OCT in routine clinical use depends upon the diagnostic sensitivity, biometric accuracy and reliability of the SD-OCT machines. This prospective, comparative, observational study aims to evaluate the imaging quality and diagnostic performance of two commercially available SD-OCT machines for both the anterior and posterior segment of the eye.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Normal eyes or
* Eyes with corneal disease:

Subjects that have any of the following conditions

1. Corneal dystrophy or degeneration
2. Corneal scarring
3. Corneal ulcer
4. Corneal injury
5. Keratoconus
6. Patients who had undergone corneal surgery
7. Patients with other corneal disease or - Eyes with retinal disease:

Subjects that have any of the following conditions:

1. Diabetic macular edema
2. Cystoid macular edema
3. Age related macular degeneration
4. Retinal vascular disorders (e.g. retinal artery occlusion)
5. Epiretinal membrane
6. Choroidal nevus
7. Macular hole
8. Patients who had undergone retinal surgery
9. Patients with other retinal disease or

   * Eyes with glaucoma
   * Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.

AND

- Written informed consent prior to recruitment

Exclusion Criteria:

Any of the following will exclude a subject from the study:

* Patients who are not able to cooperate or with insufficient ability to fixate (tremor, nystagmus)
* Pregnancy (pregnancy test will be taken in women of reproductive age before enrolment into the trial)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 eyes of 100 patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity as the proportion of anatomical structures that are detectable with the two instruments | 6 months
  Anatomical structures include e.g. sublayers of the cornea, sublayers of the retina, retinal vessels etc.

SECONDARY OUTCOMES:
Corneal sublayer thickness (µm) and retinal sublayer thickness (µm) obtained with the two study instruments | 6 months
  Comparability is analyzed between various biometric values obtained with the two instruments and typical indices of comparability are produced (e.g. intraclass correlation coefficient)
Corneal sublayer thickness and retinal sublayer thickness obtained with the two study instruments | 6 months
  Repeatability for various biometric values obtained with the two instruments is analyzed and typical indices of repeatability are produced (e.g. coefficient of variation)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Principal Investigator — AKh Linz, Augenabteilung
Locations (1):
- AKh Linz, Linz, Upper Austria, Austria

REFERENCES:
- [Derived] Luft N, Ring MH, Dirisamer M, Mursch-Edlmayr AS, Kreutzer TC, Pretzl J, Bolz M, Priglinger SG. Corneal Epithelial Remodeling Induced by Small Incision Lenticule Extraction (SMILE). Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT176-83. doi: 10.1167/iovs.15-18879. PMID 27409470